CLINICAL TRIAL: NCT04899375
Title: The Acute Effect of Tissue Flossing on Pain,Function,and Perception of Movement
Brief Title: Effect of Tissue Flossing on Pain,Function and Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Principal Investigator, Peter Douris, Professor, New York Institute of Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NewYorkIT
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Elbow Tendinopathy
Keywords: Floss band; Tissue flossing; Physical therapy; Compression
MeSH Terms: conditions — Elbow Tendinopathy

STUDY DESIGN:
Intervention Model Description: Randomized Crossover Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One group taking part in 2 separate conditions (Experimental): Subjects will be randomly assigned to either group A or B. Session 1 will serve to familiarize all participants with the battery of tests including the 100 mm VAS, Short-form Mcgill Pain Questionnaire (SF-MPQ), Likert perception scale adapted from Kiefer et al. (2017), algometry, manual muscle testing, assessed via hand-held dynamometer (HHD), and grip strength assessed via hydraulic hand dynamometer; subjects will also be instructed in the AROM protocol. Familiarization will be conducted a minimum of 24 hours prior to the first condition. There will be a minimum washout period of 1 week to reduce both order and carry-over effects. Only the principal investigator will be abreast to the order of intervention, sufficiently blinding the raters. Prior to each trial, participants will be instructed to refrain from resistance training for a minimum of 48 hours and to abstain from the use of stimulants or analgesic medication for a minimum of 6 hours prior to reporting to the lab.
  Interventions: Device: Floss band; Device: ACE bandage

INTERVENTIONS:
Device: Floss band — Tissue-flossing, is the use of an elastic band to provide compression on soft-tissue and joints whilst performing active and, or passive range of motion.
Device: ACE bandage — An ACE bandage is a cloth wrap used to provide compression

SUMMARY:
The purpose of the current investigation is to examine the effect of tissue-flossing on upper extremity, pain, strength and functional performance in subjects with musculoskeletal-related complaints of pain surrounding the elbow complex

DETAILED DESCRIPTION:
Tissue-flossing, is the use of an elastic band to provide compression on soft-tissue and joints whilst performing active and, or passive range of motion. This modality represents a contemporary strategy that has not been fully investigated with respect to performance-enhancement and rehabilitative utility.1-5 This approach was popularized by Starrett et al.(2013) with the introduction of floss-band compression for the improvement of joint specific range of motion (ROM).6 Floss bands (7'x2") are applied to site-specific muscle groups and, or joints with treatment typically lasting 1 to 3 minutes. Initial support has favored anecdote, though has a growing body of support, and carries a postulated mechanism relative to deep-tissue compression and/or reperfusion of blood.1 Despite minimal empirical evidence, this modality has gained popularity in both the sport and rehabilitation fields.1-5 There appears to be a gap in the knowledge in respect to the effectiveness of tissue-flossing Initial investigations demonstrate positive effects on ROM, jump-performance, pain, function and strength in athletic populations.1-5 Driller et al. (2017) utilized a tissue-floss technique at the ankle, to provide compression and partial vascular occlusion in recreational athletes. Performance metrics were measured for weight-bearing lunge test (WBLT), dorsi- (DF) and plantar-flexion (PF) ROM and single-leg vertical jump test for both height and velocity. The data collected from this study revealed significant improvements (p<0.01), albeit a small effect size, across all performance variables.1 Subsequently, Driller et al. (2017) investigated the time-course of tissue-flossing at the ankle, in recreational athletes.2 Performance metrics in this investigation included WBLT, counter-movement jump and 15m sprint test. Significant improvements (p<0.05) were seen, following tissue-flossing, in WBLT at all time-points, indicating a potential utility for up to 45-minutes following application.

Along with a potential performance benefit, case-studies3, 4 have presented tissue-flossing as an adjunct to conventional physical therapy. Borda et al. (2016) demonstrated efficacy in a single subject with diagnosed chronic, left Achilles tendinopathy.3 The subject (age 14), a female athlete, presented, following a 6-week course of physical therapy, with posterior ankle pain, visual analog scale (VAS) 8/10, and impaired lower extremity function, 66/80, determined by the Lower Extremity Function Scale (LEFS). Following the intervention, the patient reported a VAS of 0/10 and scored a 79/80 on the LEFS. Additionally, Arce-Esquivel et al. (2018) demonstrated effective use, in a single subject case-report, for the treatment of functional deficits and pain, associated with Keinböck's disease.4 Following 6-weeks of treatment, the patient's Wrist Hand Disability Index (WHDI) score had increased 45% from 3.3 (week 1) to 4.8 (week 6) and pain had decreased 88%, from 5.8cm/10cm (week 1) to 0.7cm/10cm (week 6). More recently, Brandenburg et al. (2018) examined the effect of tissue-flossing on imposed delayed-onset muscle soreness (DOMS) in the upper extremity. DOMS is defined as a functional muscle disorder that results from overexertion.8 Commonly, DOMS results in peak symptoms 48-72 hours post-exercise and reflects muscular pain, edema, decreased strength, power and ROM, with a concurrent neuromuscular deficit to the affected area.9-12 The investigation7 collected pain scores, via 10 cm VAS, at both 24- and 48-hours. Findings demonstrate significant improvement at both 24- (p=0.036) and 48-hours (p=0.035). The aggregate of these data suggest that tissue-flossing may be a viable supplement to clinical management of some musculoskeletal disorders. However, further research including controlled clinical trials and longitudinal observations, is warranted to further elucidate quantifiable functional outcomes and clinical application strategies associated with this modality.

In athletes, the upper extremity, specifically the elbow complex, is subject to an array of injurious processes.13 Patients often report local pain, edema, decreased strength, power and ROM, as well as, neuromuscular deficits.13,14 Manual therapy and compressive, counterforce orthoses are commonly used interventions in the non-surgical management of musculoskeletal ailments experienced at the elbow; following treatment patients report improved pain, functional performance and grip-strength.17,18 It is hypothesized that the proposed mechanisms of action, associated with tissue-flossing, may be beneficial as a cost-effective adjunct to conventional therapeutic exercise. Thus, the aim of the current investigation is to examine the effect of tissue-flossing on upper extremity functional performance in subjects with musculoskeletal-related complaints of pain surrounding the elbow complex.

ELIGIBILITY:
Inclusion Criteria:

* Elbow pain ≥1 month, VAS ≥3/10 (+) Tenderness to palpation (TTP) 1-3/4

Exclusion Criteria:

* Any condition that contraindicates the use of peripheral compression TTP >3/4

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-05-23 (Actual)

PRIMARY OUTCOMES:
VAS Pain Scale | 1 minute
  The 100 millimeter VAS is a commonly employed self-completed scale for the assessment of pain in adults. The scale is scored using a ruler, by measuring the distance in millimetres, along a 100 millimetres line, from the anchor marked "no pain".
SF-MPQ 2 | I minute
  The SF-MPQ 2 is a shorter version of the original McGill Pain Questionnaire. It is a multidimensional measure of pain, consisting of 2 subscales, one for sensory change and one for affective change.
Likert Perception Scale | I minute
  The Likert perception scale is the measurement of the subject's perception of change following the intervention.
Algometry | 3 minutes
  Algometry is the assessment of load-dependent tenderness at a specific anatomical site.
Hand held Dynamometry | 3 minutes
  HHD is a clinical tool for assessing isometric strength
Grip Strength | 3 minutes
  The assessment of hand and grip strength is a useful measure for clinicians in determining functional status.

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Douris, EdD, Principal Investigator — New York Institute of Technology
Locations (1):
- New York Institute of Technology, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Result] Driller M, Mackay K, Mills B, Tavares F. Tissue flossing on ankle range of motion, jump and sprint performance: A follow-up study. Phys Ther Sport. 2017 Nov;28:29-33. doi: 10.1016/j.ptsp.2017.08.081. Epub 2017 Aug 24. PMID 28950149
- [Result] Borda J, Selhorst M. The use of compression tack and flossing along with lacrosse ball massage to treat chronic Achilles tendinopathy in an adolescent athlete: a case report. J Man Manip Ther. 2017 Feb;25(1):57-61. doi: 10.1080/10669817.2016.1159403. Epub 2016 May 30. PMID 28855793
- [Result] Arce-Esquivel AA, Cage SA, Warner BJ, Stevenson P. Flossing bands to treat keinböck's disease in a collegiate men's basketball player: a case report. International Physical Medicine & Rehabilitation Journal. 2018;3(2).
- [Result] Kiefer BN, Lemarr KE, Enriquez CC, Tivener KA, Daniel T. A Pilot Study: Perceptual Effects of the Voodoo Floss Band on Glenohumeral Flexibility. International Journal of Athletic Therapy and Training. 2017;22(4):29-33.